CLINICAL TRIAL: NCT04867083
Title: Randomized, Open-label and Multicentric Trial Evaluating the Non-inferiority of Antiretroviral Dual Therapy Taken 4 Consecutive Days Per Week Versus Antiretroviral Dual Therapy 7/7 Days Per Week in HIV-1 Infected Patients With Controlled Viral Load Under Antiretroviral Dual Therapy
Brief Title: Dual Therapy in HIV Patients in 4 Days a Week Versus 7 Days a Week
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 177 DUETTO; 2020-003951-13 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections
Keywords: bitherapy; treatment discontinution; 4 days per week
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, prospective, randomized trial in 2 parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: 4 days/7 (Experimental): 4 days/7 Patients included in this arm will take their ARV treatment 4 consecutive days per week during 48 weeks.
  Interventions: Drug: ARV bitherapie
- Arm 2: 7 days/7 (Active Comparator): Patients included in this arm will take their ARV treatment 7 days per week during 48 weeks
  Interventions: Drug: ARV bitherapie

INTERVENTIONS:
Drug: ARV bitherapie — 1. Dolutégravir 50mg / Lamivudine 300mg per day
  2. Dolutégravir 50mg / Rilpivirine 25mg per day
  3. Darunavir/r 800mg/100mg / Lamivudine 300mg per day

SUMMARY:
The trial is an open-label, multicenter, prospective, randomized trial in 2 parallel groups, evaluating at W48 the non inferiority of antiretroviral dual therapy taken 4 consecutive days per week versus antiretroviral dual therapy 7/7 days per week in HIV-1 infected patients with controlled viral load under antiretroviral dual therapy.

DETAILED DESCRIPTION:
Open-label, multicenter, prospective, randomized trial in 2 parallel groups, evaluating at W48 the non-inferiority of antiretroviral dual therapy taken 4 consecutive days a week versus dual therapy taken 7 days a week, in HIV infected patients with controlled viral load for at least 12 months and stable antiretroviral dual therapy since 4 months. The non-inferiority margin (delta) is 5%. The randomization will be stratified according to the family of the dual therapy at the moment of the inclusion and according to the participation of the substudy or not.

The sample size calculation assumes that the true difference in efficacy between the two arms is zero and that the overall response rate is 97% at week 48. A total of 440 patients (220 per arm) is required to provide 80% power to demonstrate non-inferior efficacy for the 4/7 strategy, compared to the daily dual therapy (7/7), with a two-sided significance level of 5% and a non-inferiority margin (delta) of -5%.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, coinfection HIV-1/HIV-2 possible
* Age≥18 years old
* Current dual therapy unchanged for the last 6 months with Dolutegravir/ Lamivudine or Dolutegravir / Rilpivirine or Darunavir/r / Lamivudine
* If a genotype is available in the patient medical history; virus must be susceptible to all on going dual therapy. If no ARN genotype available, the patients can be included in the study
* Viral load (VL) < 50 c/mL in the past twelve months, with at least 3 VL measurements including screening; only one blip < 200 c/mL is authorized in the 6-12 previous months
* CD4 T cells > 250/mm3 at W-4
* Estimated glomerular filtration rate > 60 mL/min (CKD-EPI method)
* AST et ALT < 3N
* Haemoglobin > 10 g/dL
* Platelets > 100 000/mm3
* For women of childbearing age, negative pregnancy plasmatic test at W-4 and agree to use efficacy contraception during the study
* Commitment to use condom prevention and protection during sexual intercourse for the duration of the trial.
* Social security system coverage (including State Medical Aid-AME, if EC approves it)
* Informed consent form signed

Exclusion Criteria:

* Infection by HIV-2
* Chronic and active Viral B Hepatitis with positive antigen HBs
* Chronic and active Viral C Hepatitis with treatment expected in the next 48 weeks
* Concomitant treatment using interferon, interleukins, any other immune-therapy or chemotherapy, antivitamin K+ with co-treatment by booster
* Concomitant prophylactic or curative treatment for an opportunistic infection
* All conditions (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with study protocol compliance, observance and/or study treatment tolerance
* Pregnant or breast feeding women
* Subjects under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with virological failure at Week 48. | Week 48
  The virological failure is defined by 2 successive viral loads >50 c/mL at 2 to 4 weeks apart or a viral load > 50 c/ml with a definitive stop of the study follow-up or the study strategy

SECONDARY OUTCOMES:
Proportion of participants with therapeutic success until Week 48 | Week 48
Percentage of participants with at least one episode of "blip" | Week 0 to Week48
  viral load >50 copies/mL followed by a control value ≤ 50 cp/mL
Percentage of participants with a viral load signal detected | Week 0 to Week 48
Evolution of ultrasensitive viral load and total DNA in the PBMC at W0 and W48 | Week 0 and Week 48
  immuno-virological sub-study
Proportion of participants with acquisition of drugs resistance mutations in case of virological failure detected by Sanger and by NGS | Week 0 to Week 48
Description of selected mutations at the virological failure | Week 0 to Week 48
Frequency of minority resistant variants archived in DNA at W0 and their impact on virological failure (2 consecutive VL> 50 copies / mL) and on the acquisition of drugs resistance mutations | Week 0
Frequency of grade 3 or more adverse events, adverse effects, drug-modifying adverse events, drug-related adverse events and serious adverse events (SAE) | Week 0 to Week 48
Evolution of T CD4 and CD8 cells count, and CD4/CD8 ratio | Week-4 to Week 48
Evolution of fasting metabolic parameters (total cholesterol total, LDL-C, HDL-C, Triglycerides and glycemia) until W0 and W48 | Week 0 to Week 48
Evolution of weight between Week 0 and Week 48 | Week 0 and Week 48
Evolution of inflammation serum parameters | Week 0 to Week 24 and Week 48
  immuno-virological sub-study- (sCD14, sCD163, IP-10, CRPus, IL-6, D-dimers, sTNFR1, sTNFR2) from W0 to W24 and W48
Evolution of semen viral load at Week 0, Week 24 and Week 48 | Week 0-Week 24 and Week 48
  Sub-study
Description and comparison of plasmatic concentrations of antiretroviral agents between the 2 groups at ON and OFF period | Week 0-Week 8-Week 24-Week 48
Evaluation of the adherence by self-reported questionnaire | At Week 0, Week 8, Week 24, Week 36 and Week 48-the evaluation will be done after analysis of all the points
Evolution of the quality of life by self-reported questionnaire | Week-4 to Week 48-the evaluation will be done after analysis of all the points

CONTACTS AND LOCATIONS:
Overall Officials: Roland LANDMAN, Principal Investigator — Hôpital BICHAT
Locations (38):
- France (37):
  - Hôpital Louis Pasteur/Service des Maladies Infectieuses, Chartres, Le Coudray
  - Centre hospitalier Victor Dupouy/Service d'Hématologie-Unité d'Immunologie, Argenteuil
  - Hôpital Avicenne/Service des Maladies Infectieuses et tropicales, Bobigny
  - Hôpital Saint André/Service HDJ Maladies Infectieuses, Bordeaux
  - Hôpital Pellegrin/Service des Maladies Infectieuses et Tropicales, Bordeaux
  - Hôpital Côte de Nacre/Service des Maladies Infectieuses, Caen
  - Hôpital Antoine Béclère/Service d'Immunologie Clinique et Médecine Interne, Clamart
  - Centre Hospitalier Sud-Francilien/Service d'Hématologie, Corbeil-Essonnes
  - Hôpital François Mitterrand/Service des Maladies Infectieuses, Dijon
  - Hôpital Raymond Poincaré/Service des Maladies Infectieuses, Garches
  - CHD de La Roche sur Yon/Service de Médecine Interne, La Roche-sur-Yon
  - Hôpital Franco-Britannique-Fondation Cognacq-Jay, Levallois-Perret
  - CHU Dupuytren 1/Service des Maladies Infectieuses et Tropicales, Limoges
  - Hôpital de la Croix Rousse/Service des Maladies Infectieuses, Lyon
  - Hôpital Sainte Marguerite/Service d'Immuno-Hématologie Clinique, Marseille
  - Hôpital Européen/Consultation de Médecine Interne et Maladies Infectieuses, Marseille
  - Hôpital Gui de Chauliac/Service des Maladies Infectieuses, Montpellier
  - Hôpital de l'Hôtel Dieu/Service des Maladies Infectieuses, Nantes
  - Hôpital de l'Archet/Service des Maladies Infectieuses, Nice
  - Hôpital Bichat/Service des Maladies Infectieuses, Paris
  - Hôpital Hôtel Dieu/Service d'Immunologie Clinique, Paris
  - Hôpital Hôtel Dieu/Unité fonctionnelle de Pathologie Infectieuse, Paris
  - Hôpital Lariboisière/Service de Médecine Interne, Paris
  - Hôpital Saint Louis/Service des Maladies Infectieuses, Paris
  - Hôpital Saint Antoine/Service des Maladies Infectieuses, Paris
  - Hôpital Pitié-Salpêtrière/Service des Maladies Infectieuses, Paris
  - Hôpital Necker/Service des Maladies Infectieuses, Paris
  - Hôpital Tenon/Service des Maladies Infectieuses, Paris
  - Centre hospitalier de Poissy/Service des Maladies Infectieuses, Poissy
  - Centre Hospitalier René Dubos/Service de Dermatologie, Pontoise
  - Hôpital Robert DEBRE/Service des maladies infectieuses, Reims
  - Hôpital Delafontaine/Service des Maladies Infectieuses, Saint-Denis
  - Hôpital Civil/Service Le Trait D'union UF 2066, Strasbourg
  - Hôpital Foch/Service de Médecine Interne, Suresnes
  - Hôpital Purpan/Service des Maladies Infectieuses, Toulouse
  - Hôpital Gustave Dron/Service des Maladies Infectieuses, Tourcoing
  - Hôpital Bretonneau/Service des Maladies Infectieuses, Tours
- Hôpital Pierre Zobda-Quitman/Service de Médecine Interne, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer M, Hafner R, Schneider C, Trkola A, Joos B, Joller H, Hirschel B, Weber R, Gunthard HF; Swiss HIV Cohort Study. HIV RNA in plasma rebounds within days during structured treatment interruptions. AIDS. 2003 Jan 24;17(2):195-9. doi: 10.1097/00002030-200301240-00009. PMID 12545079
- [Background] Vergis EN, Paterson DL, Wagener MM, Swindells S, Singh N. Dyslipidaemia in HIV-infected patients: association with adherence to potent antiretroviral therapy. Int J STD AIDS. 2001 Jul;12(7):463-8. doi: 10.1258/0956462011923507. PMID 11394983
- [Background] Magalhaes MG, Greenberg B, Hansen H, Glick M. Comorbidities in older patients with HIV: a retrospective study. J Am Dent Assoc. 2007 Nov;138(11):1468-75. doi: 10.14219/jada.archive.2007.0083. PMID 17974644
- [Background] Ananworanich J, Nuesch R, Cote HC, Kerr SJ, Hill A, Jupimai T, Laopraynak N, Saenawat S, Ruxrungtham K, Hirschel B. Changes in metabolic toxicity after switching from stavudine/didanosine to tenofovir/lamivudine--a Staccato trial substudy. J Antimicrob Chemother. 2008 Jun;61(6):1340-3. doi: 10.1093/jac/dkn097. Epub 2008 Mar 12. PMID 18339636
- [Background] Ferry JA, Sohani AR, Longtine JA, Schwartz RA, Harris NL. HHV8-positive, EBV-positive Hodgkin lymphoma-like large B-cell lymphoma and HHV8-positive intravascular large B-cell lymphoma. Mod Pathol. 2009 May;22(5):618-26. doi: 10.1038/modpathol.2009.36. Epub 2009 Mar 13. PMID 19287457
- [Background] Ho JE, Hsue PY. Cardiovascular manifestations of HIV infection. Heart. 2009 Jul;95(14):1193-202. doi: 10.1136/hrt.2008.161463. No abstract available. PMID 19564432
- [Background] Edelman EJ, Gordon KS, Glover J, McNicholl IR, Fiellin DA, Justice AC. The next therapeutic challenge in HIV: polypharmacy. Drugs Aging. 2013 Aug;30(8):613-28. doi: 10.1007/s40266-013-0093-9. PMID 23740523
- [Background] Flandre P, Raffi F, Descamps D, Calvez V, Peytavin G, Meiffredy V, Harel M, Hazebrouck S, Pialoux G, Aboulker JP, Brun Vezinet F. Final analysis of the Trilege induction-maintenance trial: results at 18 months. AIDS. 2002 Mar 8;16(4):561-8. doi: 10.1097/00002030-200203080-00007. PMID 11872999
- [Background] Bowersox J. ACTG 343: three drugs better than two for maintaining HIV suppression. NIAID AIDS Agenda. 1998 Mar:1-2, 10-1. PMID 11365088
- [Background] Arribas JR, Girard PM, Landman R, Pich J, Mallolas J, Martinez-Rebollar M, Zamora FX, Estrada V, Crespo M, Podzamczer D, Portilla J, Dronda F, Iribarren JA, Domingo P, Pulido F, Montero M, Knobel H, Cabie A, Weiss L, Gatell JM; OLE/RIS-EST13 Study Group. Dual treatment with lopinavir-ritonavir plus lamivudine versus triple treatment with lopinavir-ritonavir plus lamivudine or emtricitabine and a second nucleos(t)ide reverse transcriptase inhibitor for maintenance of HIV-1 viral suppression (OLE): a randomised, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Jul;15(7):785-92. doi: 10.1016/S1473-3099(15)00096-1. Epub 2015 Jun 7. Erratum In: Lancet Infect Dis. 2015 Aug;15(8):875. doi: 10.1016/S1473-3099(15)00112-7. PMID 26062880
- [Background] Perez-Molina JA, Rubio R, Rivero A, Pasquau J, Suarez-Lozano I, Riera M, Estebanez M, Palacios R, Sanz-Moreno J, Troya J, Marino A, Antela A, Navarro J, Esteban H, Moreno S; GeSIDA 7011 Study Group. Simplification to dual therapy (atazanavir/ritonavir + lamivudine) versus standard triple therapy [atazanavir/ritonavir + two nucleos(t)ides] in virologically stable patients on antiretroviral therapy: 96 week results from an open-label, non-inferiority, randomized clinical trial (SALT study). J Antimicrob Chemother. 2017 Jan;72(1):246-253. doi: 10.1093/jac/dkw379. Epub 2016 Sep 13. PMID 27629070
- [Background] Di Giambenedetto S, Fabbiani M, Quiros Roldan E, Latini A, D'Ettorre G, Antinori A, Castagna A, Orofino G, Francisci D, Chinello P, Madeddu G, Grima P, Rusconi S, Di Pietro M, Mondi A, Ciccarelli N, Borghetti A, Foca E, Colafigli M, De Luca A, Cauda R; Atlas-M Study Group. Treatment simplification to atazanavir/ritonavir + lamivudine versus maintenance of atazanavir/ritonavir + two NRTIs in virologically suppressed HIV-1-infected patients: 48 week results from a randomized trial (ATLAS-M). J Antimicrob Chemother. 2017 Apr 1;72(4):1163-1171. doi: 10.1093/jac/dkw557. PMID 28093483
- [Background] Pulido F, Ribera E, Lagarde M, Perez-Valero I, Palacios R, Iribarren JA, Payeras A, Domingo P, Sanz J, Cervero M, Curran A, Rodriguez-Gomez FJ, Tellez MJ, Ryan P, Barrufet P, Knobel H, Rivero A, Alejos B, Yllescas M, Arribas JR; DUAL-GESIDA-8014-RIS-EST45 Study Group. Dual Therapy With Darunavir and Ritonavir Plus Lamivudine vs Triple Therapy With Darunavir and Ritonavir Plus Tenofovir Disoproxil Fumarate and Emtricitabine or Abacavir and Lamivudine for Maintenance of Human Immunodeficiency Virus Type 1 Viral Suppression: Randomized, Open-Label, Noninferiority DUAL-GESIDA 8014-RIS-EST45 Trial. Clin Infect Dis. 2017 Nov 29;65(12):2112-2118. doi: 10.1093/cid/cix734. PMID 29020293
- [Background] Llibre JM, Hung CC, Brinson C, Castelli F, Girard PM, Kahl LP, Blair EA, Angelis K, Wynne B, Vandermeulen K, Underwood M, Smith K, Gartland M, Aboud M. Efficacy, safety, and tolerability of dolutegravir-rilpivirine for the maintenance of virological suppression in adults with HIV-1: phase 3, randomised, non-inferiority SWORD-1 and SWORD-2 studies. Lancet. 2018 Mar 3;391(10123):839-849. doi: 10.1016/S0140-6736(17)33095-7. Epub 2018 Jan 6. PMID 29310899
- [Background] Katlama C, Assoumou L, Valantin MA, Soulie C, Martinez E, Beniguel L, Bouchaud O, Raffi F, Molina JM, Fellahi S, Peytavin G, Marcelin AG, Kolta S, Capeau J, Gibowski S, Cardon F, Reynes J, Costagliola D; members of the ANRS 163 ETRAL study. Dual therapy combining raltegravir with etravirine maintains a high level of viral suppression over 96 weeks in long-term experienced HIV-infected individuals over 45 years on a PI-based regimen: results from the Phase II ANRS 163 ETRAL study. J Antimicrob Chemother. 2019 Sep 1;74(9):2742-2751. doi: 10.1093/jac/dkz224. PMID 31269208
- [Background] Joly V, Burdet C, Landman R, Vigan M, Charpentier C, Katlama C, Cabie A, Benalycherif A, Peytavin G, Yeni P, Mentre F, Argoud AL, Amri I, Descamps D, Yazdanpanah Y; LAMIDOL Study Group. Dolutegravir and lamivudine maintenance therapy in HIV-1 virologically suppressed patients: results of the ANRS 167 trial (LAMIDOL). J Antimicrob Chemother. 2019 Mar 1;74(3):739-745. doi: 10.1093/jac/dky467. PMID 30476165
- [Background] Taiwo BO, Marconi VC, Berzins B, Moser CB, Nyaku AN, Fichtenbaum CJ, Benson CA, Wilkin T, Koletar SL, Colasanti J, Acosta EP, Li JZ, Sax PE. Dolutegravir Plus Lamivudine Maintains Human Immunodeficiency Virus-1 Suppression Through Week 48 in a Pilot Randomized Trial. Clin Infect Dis. 2018 May 17;66(11):1794-1797. doi: 10.1093/cid/cix1131. PMID 29293895
- [Background] van Wyk J, Ajana F, Bisshop F, De Wit S, Osiyemi O, Portilla Sogorb J, Routy JP, Wyen C, Ait-Khaled M, Nascimento MC, Pappa KA, Wang R, Wright J, Tenorio AR, Wynne B, Aboud M, Gartland MJ, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose 2-Drug Regimen vs Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Phase 3, Randomized, Noninferiority TANGO Study. Clin Infect Dis. 2020 Nov 5;71(8):1920-1929. doi: 10.1093/cid/ciz1243. PMID 31905383
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Dybul M, Chun TW, Yoder C, Hidalgo B, Belson M, Hertogs K, Larder B, Dewar RL, Fox CH, Hallahan CW, Justement JS, Migueles SA, Metcalf JA, Davey RT, Daucher M, Pandya P, Baseler M, Ward DJ, Fauci AS. Short-cycle structured intermittent treatment of chronic HIV infection with highly active antiretroviral therapy: effects on virologic, immunologic, and toxicity parameters. Proc Natl Acad Sci U S A. 2001 Dec 18;98(26):15161-6. doi: 10.1073/pnas.261568398. Epub 2001 Dec 4. PMID 11734634
- [Background] Dybul M, Nies-Kraske E, Dewar R, Maldarelli F, Hallahan CW, Daucher M, Piscitelli SC, Ehler L, Weigand A, Palmer S, Metcalf JA, Davey RT, Rock Kress DM, Powers A, Beck I, Frenkel L, Baseler M, Coffin J, Fauci AS. A proof-of-concept study of short-cycle intermittent antiretroviral therapy with a once-daily regimen of didanosine, lamivudine, and efavirenz for the treatment of chronic HIV infection. J Infect Dis. 2004 Jun 1;189(11):1974-82. doi: 10.1086/386344. Epub 2004 May 10. PMID 15143462
- [Background] Cohen CJ, Colson AE, Sheble-Hall AG, McLaughlin KA, Morse GD. Pilot study of a novel short-cycle antiretroviral treatment interruption strategy: 48-week results of the five-days-on, two-days-off (FOTO) study. HIV Clin Trials. 2007 Jan-Feb;8(1):19-23. doi: 10.1310/hct0801-19. PMID 17434845
- [Background] Cohen C, Colson A, Pierone G. The FOTO study: Twenty-Four week results support the safety of a two day break on efavirenz-based antiretroviral therapy. Presented at: Ninth International Congress on Drug Therapy in HIV Infection; November 8-13, 2008; Glasgow, UK
- [Background] Cohen C, Colson A, Pierone G, et al. The FOTO study: The 48 week extension to assess durability of the strategy of taking efavirenz, tenofovir and emtricitabine Five days On, Two days Off (FOTO) each week in virologically suppressed patients. Presented at: Fifth International AIDS Society Conference on HIV Pathogenesis, Treatment, and Prevention; July 19-22, 2009; Cape Town, South Africa
- [Background] Reynolds SJ, Kityo C, Hallahan CW, Kabuye G, Atwiine D, Mbamanya F, Ssali F, Dewar R, Daucher M, Davey RT Jr, Mugyenyi P, Fauci AS, Quinn TC, Dybul MR. A randomized, controlled, trial of short cycle intermittent compared to continuous antiretroviral therapy for the treatment of HIV infection in Uganda. PLoS One. 2010 Apr 22;5(4):e10307. doi: 10.1371/journal.pone.0010307. PMID 20442758
- [Background] Leibowitch J, Mathez D, de Truchis P, Ledu D, Melchior JC, Carcelain G, Izopet J, Perronne C, David JR. Four days a week or less on appropriate anti-HIV drug combinations provided long-term optimal maintenance in 94 patients: the ICCARRE project. FASEB J. 2015 Jun;29(6):2223-34. doi: 10.1096/fj.14-260315. Epub 2015 Apr 1. PMID 25833895
- [Background] BREATHER (PENTA 16) Trial Group. Weekends-off efavirenz-based antiretroviral therapy in HIV-infected children, adolescents, and young adults (BREATHER): a randomised, open-label, non-inferiority, phase 2/3 trial. Lancet HIV. 2016 Sep;3(9):e421-e430. doi: 10.1016/S2352-3018(16)30054-6. Epub 2016 Jun 20. PMID 27562743
- [Background] de Truchis P, Assoumou L, Landman R, Mathez D, Le Du D, Bellet J, Amat K, Katlama C, Gras G, Bouchaud O, Duracinsky M, Abe E, Alvarez JC, Izopet J, Saillard J, Melchior JC, Leibowitch J, Costagliola D, Girard PM, Perronne C; ANRS 162-4D Study Group. Four-days-a-week antiretroviral maintenance therapy in virologically controlled HIV-1-infected adults: the ANRS 162-4D trial. J Antimicrob Chemother. 2018 Mar 1;73(3):738-747. doi: 10.1093/jac/dkx434. PMID 29186458
- [Background] R. Landman, P. De Truchis, L. Assoumou, S. Lambert, K. Amat, J. Bellet, B. Lefebvre, C. Allavena, C. Katlama, Y. Yazdanpanah, J.-M. Molina, A. Gelley, S. Gibowski, J.-C. Alvarez, L. Morand-Joubert, D. Costagliola, P.-M. Girard, ANRS 170 QUATUOR study group -ANRS 170 QUATUOR 4/7 days maintenance strategy in antiretroviral treated adults with HIV-1 infection: an open randomised parallel non-inferiority phase III trial Abstract IAS2019 WEAB0406LB
- [Background] Parienti JJ, Das-Douglas M, Massari V, Guzman D, Deeks SG, Verdon R, Bangsberg DR. Not all missed doses are the same: sustained NNRTI treatment interruptions predict HIV rebound at low-to-moderate adherence levels. PLoS One. 2008 Jul 30;3(7):e2783. doi: 10.1371/journal.pone.0002783. PMID 18665246
- [Background] Pogany K, van Valkengoed IG, Prins JM, Nieuwkerk PT, van der Ende I, Kauffmann RH, Kroon FP, Verbon A, Nievaard MF, Lange JM, Brinkman K. Effects of active treatment discontinuation in patients with a CD4+ T-cell nadir greater than 350 cells/mm3: 48-week Treatment Interruption in Early Starters Netherlands Study (TRIESTAN). J Acquir Immune Defic Syndr. 2007 Apr 1;44(4):395-400. doi: 10.1097/QAI.0b013e31802f83bc. PMID 17195761
- [Background] Zehnacker L, Abe E, Mathez D, Alvarez JC, Leibowitch J, Azoulay S. Plasma and Intracellular Antiretroviral Concentrations in HIV-Infected Patients under Short Cycles of Antiretroviral Therapy. AIDS Res Treat. 2014;2014:724958. doi: 10.1155/2014/724958. Epub 2014 Nov 9. PMID 25431661